CLINICAL TRIAL: NCT02800824
Title: Bioequivalence Study of Budesonide Rectal Aerosol Foam and Uceris® Rectal Aerosol Foam
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Padagis LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: PRG-NY-16-007
Record Dates: First submitted 2016-06-07; First posted 2016-06-15 (Estimated); Last update posted 2022-01-13 (Actual); Status verified 2021-12

CONDITIONS: Healthy
MeSH Terms: interventions — Budesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Budesonide rectal foam (Experimental)
  Interventions: Drug: Budesonide
- Uceris rectal foam (Active Comparator)
  Interventions: Drug: Uceris

INTERVENTIONS:
Drug: Budesonide
  Arms: Budesonide rectal foam
Drug: Uceris
  Arms: Uceris rectal foam

SUMMARY:
To evaluate the bioequivalence between the Test Product Budesonide rectal aerosol foam and Reference Product Uceris® rectal aerosol foam after a single-dose in healthy subjects

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, non-smoking, male and female subjects, 18 years of age or over.
2. No clinically significant findings in vital signs measurements or 12-lead electrocardiogram (ECG) or abnormal laboratory values.
3. Have no significant diseases.
4. Willing to use an acceptable, effective method of contraception.
5. Informed on the nature of the study and have agreed to and are able to read, review and sign all consent documents.
6. Have no clinically significant findings from a physical examination.

Exclusion Criteria:

1. Known history or presence of clinically significant neurologic, hematologic, endocrine, oncologic, pulmonary, immunologic, genitourinary, psychiatric, or cardiovascular disease or any other condition which, in the opinion of the Investigator, would jeopardize the safety of the subject or impact the validity of the study results
2. Known history or presence of hypersensitivity or idiosyncratic reaction to budesonide, any other components of the drug products, or any other drug substances with similar activity or sodium phosphate
3. History or presence or of diabetes mellitus, glaucoma or cataracts, hypertension, or osteoporosis
4. History of drug or alcohol addiction requiring treatment.
5. History of malabsorption within the last year.
6. Presence of hepatic or renal dysfunction.
7. Presence of a medical condition requiring regular medication (prescription and/or over-the-counter) with systemic absorption.
8. Positive test result for HIV, Hepatitis B surface antigen, or Hepatitis C antibody.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Primary Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma drug concentration (Cmax) | 24 hours
AUC from time 0 extrapolated to infinity (AUC0-∞) | 24 hours
AUC from time 0 to 24 hours (AUC0-24) | 24 hours

IPD SHARING:
Plan to Share IPD: No